CLINICAL TRIAL: NCT05360550
Title: A Study to Evaluate the Effect of a Contraceptive Vaginal Ring LSP- 5415 Releasing Ethinyl Estradiol Plus Etonogestrel on Ovarian Function in Healthy Adult Females
Brief Title: A Study to Evaluate the Effect of a Contraceptive Vaginal Ring LSP- 5415 on Ovarian Function in Healthy Adult Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lupin Research Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CVR-WH-202
Record Dates: First submitted 2022-01-21; First posted 2022-05-04 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy Prevention

STUDY DESIGN:
Intervention Model Description: The study will consist of two subject cohorts; Cohort #1 will consist of a total of 16 healthy women aged 18-35 years with a BMI of ≥ 18 kg/m2 to ≤ 30 kg/m2, Cohort #2 will consist of up to 10 healthy women aged 18-35 years with a BMI of > 30 kg/m2 to ≤ 35 kg/m2. The study will consist of 3 treatment cycles each consisting of a 26 day ring-insertion period followed by a 2-day ring-free period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LSP-5415 (etonogestrel/ethinyl estradiol vaginal ring) (Experimental): LSP-5415
  Interventions: Drug: LSP-5415

INTERVENTIONS:
Drug: LSP-5415 — pregnancy prevention

SUMMARY:
The primary objective of this study is to evaluate the inhibition of ovulation in Cohort #1 (Body Mass Index of ≥ 18 kg/m2 to ≤ 30 kg/m2) after contraceptive vaginal ring LSP-5415 application for 3 treatment cycles.

DETAILED DESCRIPTION:
This is an open-label study to evaluate inhibition of ovulation during treatment with LSP-5415 over a period of 3 treatment cycles (approximately 3 months) in healthy female volunteers with a documented ovulatory cycle (pre-treatment cycle). The study will consist of two subject cohorts; Cohort #1 will consist of a total of 16 healthy women aged 18-35 years with a BMI of ≥ 18 kg/m2 to ≤ 30 kg/m2, Cohort #2 will consist of up to 10 healthy women aged 18-35 years with a BMI of > 30 kg/m2 to ≤ 35 kg/m2. The study will consist of 3 treatment cycles each consisting of a 26 day ring-insertion period followed by a 2-day ring-free period.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to read and write and willing to sign Informed Consent Form prior to study participation in accordance with legal requirements.
2. Females (18 to 35 years of age, inclusive) without uncontrolled concomitant disease at the Baseline Visit.
3. Have a regular menstrual cycle that is 24-32 days in duration.
4. Cohort #1 - BMI of 18 kg/m2 to 30 kg/m2, inclusive. Cohort #2 - BMI > 30 kg/m2 to ≤ 35 kg/m2. -
5. Will not be at risk for pregnancy; subjects must agree to consistently use reliable non-hormonal contraceptive methods (spermicide-coated condoms, sterilization, male partner's sterilization via vasectomy, or sexual abstinence), or be in a same-sex relationship from screening through study completion or be surgically sterilized by bilateral tubal ligation.
6. Both ovaries and uterus must be intact, and visible on transvaginal ultrasound (TVUS) examination during screening.
7. Subjects must be in good physical and mental health as determined by vital signs, medical history and clinical examination.
8. Subjects must have a blood pressure reading in a sitting position, between 90-140 mmHg (systolic) and 50-90 mmHg (diastolic) and pulse rate between 50 and 100 bpm.
9. Be at least 3 months after a delivery or abortion.
10. Be at least six months since last progestin injection with one or more spontaneous menses.
11. Willing to abstain from vaginal products e.g., tampons, intravaginal medications etc. during the ring wear period for the study duration except water based vaginal lubricants/spermicides.

Exclusion Criteria:

1. Pregnancy, a positive serum β-hCG pregnancy test at screening or lactation.
2. Use of tobacco- or nicotine-containing products (e.g., cigarette, pipe, cigar, chewing, nicotine patch, or nicotine gum) within 6 months prior to study drug administration on Day 1 of treatment cycle 1.
3. Have a history of cervical carcinoma or other carcinomas of the vagina or vulva.
4. Subjects with abnormal pap smears that require colposcopic evaluations as defined by the fourth American Society of Colposcopy and Cervical Pathology (ASCCP) sponsored guidelines for management of cervical cancer abnormalities during the next 6 months are excluded. Subjects with abnormal pap smear and who have undergone colposcopic evaluation which has determined that a cervical procedure is not necessary during the 6 months following the colposcopy are allowed.
5. Breast cancer or other estrogen- or progestin-sensitive cancer, now or in the past.
6. History of thrombophlebitis, venous or arterial thromboembolic diseases (thrombosis, pulmonary embolism, stroke or myocardial infarction).
7. Any known severe neurological, gastrointestinal, hepatic (liver tumors, benign or malignant or liver disease) or other disease that might interfere with the intake of an investigational drug or any study condition.
8. Planned surgical procedures during the study period.
9. Clinically relevant/significant findings from serum biochemistry and hematology and HBsAg and C Virus/HlV serology as evaluated by the investigator.
10. Clinically relevant electrocardiogram (ECG) findings.
11. Anovulatory pre-treatment cycle, or no ovulation by Day 27 of the pretreatment cycle, or sonographical peculiarities concerning the ovarian status (e.g., ovarian cyst formation), that have not disappeared during the pretreatment cycle.
12. Ovarian cyst larger than 3 cm in largest dimension on TVUS that persists during the pre-treatment ovulatory cycle.
13. Additional contraindications related to the use of ethinyl estradiol (EE), or hormonal contraceptives including women with a high risk of arterial or venous thrombotic diseases. Examples include women who are known to:

    1. Have cerebrovascular disease
    2. Have coronary artery disease -
    3. Have thrombogenic valvular or thrombogenic rhythm diseases of the heart (for example, subacute bacterial endocarditis with valvular disease, or atrial fibrillation)
    4. Have inherited or acquired hypercoagulopathies
    5. Have uncontrolled hypertension
    6. Have diabetes mellitus with vascular disease
    7. Have headaches with focal neurological symptoms or migraine headaches with aura
14. History of migraine with focal neurological symptoms.
15. Known hereditary or acquired predisposition for venous and/or arterial thromboembolism (e.g., activated protein C [APC] resistance, anticardiolipin antibodies).
16. Less than 2 weeks remobilization after major surgery or prolonged immobilization.
17. Alcohol, drug, or medicine abuse, or suspicion thereof.
18. Known allergy to any ingredient of the investigational drug.
19. Use of long-acting injectable or implant hormonal therapy. A washout period of 10 months and two regular cycles is required after use of long-acting injectable contraceptive therapy (depo-medroxyprogesterone) or implant hormonal therapy prior to the pre-treatment cycle.
20. Use of hormonal or non-hormonal Intrauterine devices (IUDs) within 30 days prior to the start of the pre-treatment cycle.
21. Participation in another clinical trial at same time or within the preceding three months.
22. Subjects with a desire to become pregnant during the study.
23. Undiagnosed vaginal discharge, vaginal lesions/abnormalities or undiagnosed abnormal uterine bleeding. Subjects suspected of having a vaginal infection (e.g., chlamydia, gonococcus, yeast, trichomoniasis, or bacterial vaginosis, etc.) may be enrolled after treatment and subsequent negative test results; partner treatment is also recommended (as per treatment guidelines).
24. Regular intake or use of the following medication:

    1. any drugs that might interfere with the investigational drug.
    2. any hormonal preparation one cycle prior to the start of the pre-treatment cycle until the end of treatment cycles (except for thyroid disorders under control).
    3. any drugs known to induce liver enzymes (e.g., rifampicin, dexamethasone, barbiturates, anticonvulsants, St. John's Wort).
    4. any drugs known to inhibit CYP 3A4 (e.g. ketoconazole, verapamil, cimetidine, macrolides).
    5. any broad-spectrum antibiotics.
    6. any Hepatitis C drug combinations containing ombitasvir/paritaprevir/ritonavir, with or without dasabuvir, due to potential for ALT elevations.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Adult Females
Enrollment: 26 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in Cohort #1 with complete ovarian inhibition over 3 treatment cycles | 3 months
  The primary endpoint is the proportion of subjects in Cohort #1 with complete ovarian inhibition over the entire treatment period (3 treatment cycles). Ovarian inhibition will be assessed by rating the suppression of ovaries using the
  Hoogland score (Hoogland HJ, Skouby SO, 1993). This score is based on:
  * The follicular size assessed by transvaginal ultrasound (TVUS).
  * Endogenous hormone levels: serum Estradiol (E2), and serum Progesterone (P). A Hoogland and Skouby grade 3 and below represents ovulation inhibition

SECONDARY OUTCOMES:
Measurement of Serum level of Luteinizing Hormone (LH) | 3 months
  Serum level of Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH), E2, P
Measurement of Plasma level of Ethinyl Estradiol (EE), Etonogestrel (ENG) | 3 months
  Plasma level of Ethinyl Estradiol (EE), Etonogestrel (ENG): Blood samples will be taken at regular time points during Cycle 3 (26-day wear period).
Measurement of Samples for sex hormone-binding globulin (SHBG) | 3 months
  Samples for sex hormone-binding globulin (SHBG) will be collected preinsertion on Cycle 1, Day 1 and pre-removal on Cycle 3, Day 27.
Safety (Number of study subjects with treatment-emergent adverse events) | 3 months
  To assess the safety of LSP-5415 in healthy adult female subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Mohope, Mumbai, India